CLINICAL TRIAL: NCT05123703
Title: A Phase III Multicenter, Randomized, Double-blind, Double-dummy Study to Evaluate Safety and Efficacy of Ocrelizumab in Comparison With Fingolimod in Children and Adolescents With Relapsing-Remitting Multiple Sclerosis
Brief Title: A Study to Evaluate Safety and Efficacy of Ocrelizumab in Comparison With Fingolimod in Children and Adolescents With Relapsing-Remitting Multiple Sclerosis (RRMS)
Acronym: Operetta 2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WN42086; 2020-004128-41 (EudraCT Number); 2023-506516-40-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2021-11-16; First posted 2021-11-17 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
Keywords: pediatric Multiple Sclerosis; pediatric MS; children MS; children Multiple Sclerosis; pediatric ocrelizumab
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — ocrelizumab; Fingolimod Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ocrelizumab (Experimental): Participants will receive ocrelizumab by intravenous (IV) infusion every 24 weeks (Q24W). The first dose is given as dual infusions of half the dose of ocrelizumab on Days 1 and 15 and subsequent doses are given as single infusions of ocrelizumab Q24W. Participants will also receive a placebo of fingolimod administered as once a day (QD) capsule.
  Interventions: Drug: Ocrelizumab; Other: Fingolimod Placebo
- Fingolimod (Active Comparator): Participants will receive fingolimod orally (PO) QD as per the prescribing information provided with fingolimod. Participants will also receive a placebo of ocrelizumab administered as IV infusion on Days 1 and 15, and Q24W thereafter.
  Interventions: Other: Ocrelizumab Placebo; Drug: Fingolimod

INTERVENTIONS:
Drug: Ocrelizumab — Ocrelizumab 300 milligrams (mg) will be administered by IV infusion to participants who weigh < 35 kilograms (kg) and ocrelizumab 600 mg IV will be administered to participants who weigh ≥ 35 kg on Days 1 and 15 (half the dose, 2 weeks apart) and Q24W thereafter.
  Arms: Ocrelizumab
Other: Ocrelizumab Placebo — Ocrelizumab matching placebo will be administered by IV infusion on Day 1 and Day 15 and Q24W thereafter.
  Arms: Fingolimod
Drug: Fingolimod — Fingolimod will be administered daily as a capsule per the prescribing information (0.25 mg to participants who weigh ≤ 40 kg and 0.5 mg to participants who weigh > 40 kg).
  Arms: Fingolimod
Other: Fingolimod Placebo — Fingolimod matching placebo will be administered daily as a capsule.
  Arms: Ocrelizumab

SUMMARY:
This double-blind, double-dummy study will evaluate the safety and efficacy of ocrelizumab compared with fingolimod in children and adolescents with RRMS aged between 10 and < 18 years over a flexible duration. The double-blind period will last until after the last participant randomized has completed 24 weeks.

DETAILED DESCRIPTION:
This Phase III randomized, double-blind, double-dummy, multicenter study will evaluate the safety and efficacy of ocrelizumab administered by IV infusion every 24 weeks compared with fingolimod taken orally daily, in children and adolescents with RRMS aged between 10 and < 18 years. The study plans to enroll 171 participants in a 1:1 randomization (ocrelizumab:fingolimod), globally. This study consists of a double-blind, double dummy period in which participants will be treated with either active ocrelizumab or active fingolimod for a flexible duration. Participants who complete the double-blind period will be offered the possibility to enter an optional open-label extension (OLE) treatment period of at least 144 weeks with ocrelizumab.

ELIGIBILITY:
Inclusion Criteria:

* Body weight ≥ 25 kilograms (kg)
* Diagnosis of RRMS in accordance with the International Pediatric Multiple Sclerosis Study Group (IPMSSG) criteria for pediatric Multiple Sclerosis (MS), Version 2012, or McDonald criteria 2017
* Expanded Disability Status Scale (EDSS) at screening: 0-5.5, inclusive
* For all countries except Germany, at least one MS relapse during the previous year or two MS relapses in the previous 2 years or evidence of at least one Gd enhancing lesion on MRI within 6 months

Inclusion Criteria for Optional OLE Period:

-Participants in Group A (ocrelizumab in the double-blind period [DBP]) and Group B (fingolimod in the DBP) who, in the opinion of the investigator, may benefit from switching to ocrelizumab and who have completed the DBP with study treatment (ocrelizumab/fingolimod), may participate in the OLE period

Exclusion Criteria:

* Known presence or suspicion of other neurologic disorders that may mimic MS
* Significant uncontrolled somatic diseases, known active infection or any other significant condition that may preclude participant from participating in the study
* Participants with severe cardiac disease or significant findings on the screening Electrocardiograph (ECG)

Exclusion Criteria for Optional OLE Period:

-Participants who have discontinued the study during the DBP

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 188 (Actual)
Dates: Start 2022-05-19 (Actual); Primary Completion 2025-06-09 (Actual); Study Completion 2029-09-17 (Estimated)

PRIMARY OUTCOMES:
Annualized Relapse Rate (ARR) | Baseline up to approximately 4 years

SECONDARY OUTCOMES:
Number of New or Enlarging T2-hyperintense Lesions (T2 lesions) as Detected by Brain Magnetic Resonance Imaging (MRI) During the Double-blind Period | Baseline up to approximately 4 years
Number of New or Enlarging T2 Lesions by Week 96 | Baseline up to Week 96
ARR by Week 96 | Baseline up to Week 96
Number of T1 Gadolinium (Gd) Lesions at Week 12 | Week 12
Incidence and Severity of Adverse Events (AEs), With Severity Determined According to National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (NCI CTCAE v5.0) | Baseline up to approximately 8 years
Prevalence of Anti-drug Antibodies (ADAs) at Baseline and Incidence of ADAs During the Study | Baseline up to approximately 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (102):
- United States (13):
  - UC San Diego, La Jolla, California
  - University of California San Francisco, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Hospital, Washington D.C., District of Columbia
  - Johns Hopkins Medicine, Baltimore, Maryland
  - Boston Children's Hospital Central Pharmacy, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Cleveland Clinic, Mellen Center for Multiple Sclerosis, Cleveland, Ohio
  - The Boster Center for Multiple Sclerosis a Singlepoint Healthcare Company, Columbus, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Baylor College of Medicine/Texas Children's Hospital, Houston, Texas
  - University of Virginia Health System, Charlottesville, Virginia
- Argentina (3):
  - Hospital de Pediatría S.A.M.I.C.- Prof. Dr. Juan P. Garrahan, Ciudad de Buenos Aires
  - Clinica Universitaria Reina Fabiola, Córdoba
  - Centro de Investigaciones Médicas Tucuman, San Miguel de Tucumán
- Royal Children's Hospital Melbourne - PIN, Parkville, Victoria, Australia
- Medizinische Universität Wien, Vienna, Austria
- Belgium (3):
  - Hôpital Universitaire des Enfants Reine Fabiola, Brussels
  - Cliniques Universitaires St-Luc, Brussels
  - UZ Gent, Ghent
- Brazil (7):
  - L2 Ip - Instituto de Pesquisas Clinicas Ltda - ME, Brasília, Federal District
  - Instituto de Neurologia de Curitiba, Curitiba, Paraná
  - Universidade de Caxias do Sul - Rio Grande do Sul, Caxias do Sul, Rio Grande do Sul
  - Nucleo de Pesquisa Clinica do Rio Grande do Sul NPCR, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
  - CPQuali Pesquisa Clínica Sao Paulo, São Paulo, São Paulo
  - Inst. Da Criança- Faculdade de Medicina Usp, São Paulo
- Canada (3):
  - University of Alberta Hospital, Edmonton, Alberta
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
- Estonia (2):
  - Astra Kliinik, Tallinn
  - Tartu University Hospital, Tartu
- France (4):
  - Hospices Civils de Lyon - Hôpital Pierre Wertheimer, Bron, Rhône
  - Centre Hospitalier Universitaire de Bicêtre, Le Kremlin-Bicêtre
  - CHRU de Montpellier, Hopital Gui de Chauliac, Montpellier
  - Hopital de Hautepierre, Strasbourg
- Germany (4):
  - Vestische Kinder- und Jugendklinik Datteln, Datteln
  - Universitaetsklinikum Carl Gustav Carus an der TU Dresden, Dresden
  - Universitätsmedizin Göttingen Georg-August-Universität, Göttingen
  - Universitätsklinikum Münster, Münster
- Greece (3):
  - Eginitio University General Hospital of Athens, Athens, Attica
  - University General Hospital ''ATTIKON'' - General Hospital of West Attica H AGIA VARVARA, Chaïdári, Attica
  - St. Luke's Hospital, Thessaloniki
- Hungary (2):
  - Semmelweis Egyetem, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
- India (7):
  - Zydus Hospital, Ahmedabad, Gujarat
  - Artemis Hospital, Gurugram, Haryana
  - Sparsh Super Speciality Hospital, Bangalore North, Karnataka
  - Amrita Institute of Medical Sciences and Research Centre, Kochi, Kerala
  - Deenanath Mangeshkar Hospital & Research Centre, Pune, Maharashtra
  - All India Institute Of Medical Sciences (AIIMS), New Delhi, National Capital Territory of Delhi
  - Fortis Flight Lieutenant Rajan Dhall Hospital, New Delhi, National Capital Territory of Delhi
- Italy (7):
  - Universita? G. D'Annunzio, Chieti, Abruzzo
  - Azienda Ospedaliero-Universitaria Consorziale Pol. di Bari, Bari, Apulia
  - IRCCS Materno Infantile Burlo Garofolo - INCIPIT - PIN, Trieste, Friuli Venezia Giulia
  - Ospedale Pediatrico Bambino Gesù, Rome, Lazio
  - Azienda Ospedaliera Sant'Andrea, Rome, Lazio
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan, Lombardy
  - Azienda Ospedaliero Universitaria Policlinico Vittorio Emanuele, Catania, Sicily
- Children's Clinical University Hospital, Riga, Latvia
- Mexico (8):
  - Hospital Civil Fray Antonio Alcalde, Guadalajara, Jalisco
  - Clinstile S.A de C.V., Mexico City, Mexico CITY (federal District)
  - Grupo Médico Camino S.C., Mexico City, Mexico CITY (federal District)
  - Centro de Investigacion Clinica Chapultepec S. A. de C. V., Morelia, Michoacán
  - Iecsi S.C., Monterrey, Nuevo León
  - Neurociencias Estudios Clinicos S.C., Culiacán, Sinaloa
  - Centro para el Desarrollo de la Medicina y de Asistencia, Culiacán, Sinaloa
  - FAICIC S de R.L. de C.V, Veracruz
- Morocco (4):
  - Hassan II University Hospital, Fes
  - CHU Mohammed VI, Marrakesh
  - Centre Hospitalier Ibn Sina CHIS - Hopital des Specialites, Rabat
  - Hospital Militaire Dinstruction Mohammed V de Rabat, Rabat
- Poland (5):
  - Instytut Centrum Zdrowia Matki Polki, ?ód?
  - Uniwersyteckie Centrum Kliniczne, Gda?sk
  - Uniwersytecki Szpital Kliniczny w Poznaniu, Późna
  - Dzieci?cy Szpital Kliniczny im. Józefa Polikarpa Brudzi?skiego, Warsaw
  - Instytut Pomnik Centrum Zdrowia Dziecka, Warsaw
- Portugal (4):
  - Hospital de Braga, Braga
  - ULS de Coimbra, EPE - Hospitais da Universidade de Coimbra, Coimbra
  - Hospital Santo Antonio dos Capuchos, Lisbon
  - Centro Hospitalar Lisboa Norte, E.P.E. ? Hospital de Santa Maria, Lisbon
- Romania (2):
  - Victor Gomoiu Clinical Hospital for Children, Bucharest
  - Prof Dr Alexandru Obregia Clinical Psychiatric Hospital, Bucharest
- Serbia (4):
  - Childrens University Hospital, Belgrade
  - Clinic for Neurology and Psychiatry for Children and Youth, Belgrade
  - Mother and Child Health Care Institute of Serbia Dr Vukan Cupic, Belgrade
  - University Clinical Centre of Nis, Niš
- Spain (7):
  - Hospital Sant Joan De Deu, Esplugues de Llobregas, Barcelona
  - Hospital de Cruces, Barakaldo, Vizcaya
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario de la Princesa, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Regional Universitario Carlos Haya, Málaga
  - Hospital Universitario Virgen Macarena, Seville
- Universitäts-Kinderspital Zürich - Eleonorenstiftung, Zurich, Switzerland
- Ukraine (3):
  - Communal noncommercial enterprise of Lviv Regional Council Lviv Regional Clinical Hospital, Lviv, Kharkiv Governorate
  - Ukrainian medical rehabilitation center for children with organic lesions of the nervous system, Kyiv, KIEV Governorate
  - KZ "Dnipropetrovska oblasna dytiacha klinichna likarnia" DOR, Dnipropetrovsk, Tavria Okruha
- United Kingdom (3):
  - Addenbrookes Hospital, Cambridge
  - Royal Hospital for Children and Young People, Edinburgh
  - Great Ormond Street Hospital For Children, London

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Mar S, Valeriani M, Steinborn B, Schreiner T, Waubant E, Filippi M, Kotulska K, Mazurkiewicz-Beldzinska M, El Azzouzi B, Lin CJ, Shen YA, Kletzl H, Evershed J, Hogea A, Manlius C, Bonati U, Banwell B. Ocrelizumab dose selection for treatment of pediatric relapsing-remitting multiple sclerosis: results of the OPERETTA I study. J Neurol. 2025 Jan 15;272(2):137. doi: 10.1007/s00415-024-12879-z. PMID 39812825